CLINICAL TRIAL: NCT05061524
Title: A First-in-Human, Randomized, Double-Blind, Placebo/Active Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Following Subcutaneous Injections of YH35324 in Atopic Healthy Subjects or Subjects with Mild Allergic Diseases
Brief Title: A FIH Study of YH35324 in Atopic Healthy Subjects or Subjects with Mild Allergic Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH35324-101
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Atopic Healthy Subjects; Adult Subjects with Mild Allergic Diseases
Keywords: YH35324; GI-301; Allergic disease
MeSH Terms: interventions — Omalizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- YH35324 (Experimental): * Part A: A single dose of the YH35324 will be administered subcutaneously in 5 dose groups (0.3, 1, 3, 6, and 9 mg/kg), and a dose will be escalated in a stepwise manner from low to high doses
  * Part B: A single dose of the YH35324 will be administered subcutaneously. The dose of YH35324 will be determined after the safety, tolerability, PK, and PD data in Part A are reviewed
  Interventions: Drug: YH35324
- Placebo (Placebo Comparator): * Part A: A single dose of the Placebo will be administered subcutaneously in 5 Cohorts(Dose groups=0.3, 1, 3, 6, and 9 mg/kg), and a dose will be escalated in a stepwise manner from low to high doses
  * Part B: Placebo is not administered in Part B
  Interventions: Drug: Placebo
- Xolair® for injection (Omalizumab) (Active Comparator): * Part A: A single fixed dose of the Omalizumab 300mg will be administered subcutaneously in 4 Cohorts(Dose groups of YH35324=1, 3, 6, and 9 mg/kg)
  * Part B: A single dose of the Omalizumab 300mg will be administered subcutaneously.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: YH35324 — Subcutaneous injection of YH35324
  Arms: YH35324
Drug: Placebo — Subcutaneous injection of None of active ingredient
  Arms: Placebo
Drug: Omalizumab — Subcutaneous injection of Omalizumab
  Other Names: Xolair® for injection
  Arms: Xolair® for injection (Omalizumab)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK, and PD following subcutaneous injections of YH35324 in atopic healthy subjects or adult subjects with mild allergic diseases. Eligible subjects will be randomized to the YH35324 group, the placebo group, or the omalizumab group.

DETAILED DESCRIPTION:
YH35324 is a drug under development as a novel therapeutic agent for various IgE-mediated allergic diseases. Since YH35324 has a high binding affinity to human IgE, it prevents serum IgE from binding to receptors on mast cells and basophil, thereby inhibiting histamine release caused by degranulation when exposed to allergens Based on its non-clinical study results, this study aims to evaluate the safety, tolerability, PK, and PD following subcutaneous injections of YH35324 in atopic healthy subjects or subjects with mild allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years old, Atopic Healthy Subjects or Subjects With Mild Allergic Diseases
* Serum total IgE level of 30 to 700 IU/mL or > 700 IU/mL
* Signed the informed consent form

Exclusion Criteria:

* Hyperimmunoglobulin E syndrome or malignancy
* Positive drug screen result
* AST or ALT > 1.5 * Upper normal range
* eGFR < 60mL/min/1.73m2
* Allergy immunotherapy initiated or Administration of a live vaccine within 3 months prior to randomization
* History of participation in another clinical trial within 6 months prior to randomization

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability following single administration of YH35324 | Occurrence and severity of adverse events will be observed for 113 days after administration
  Occurrence and severity of adverse events (AEs)

SECONDARY OUTCOMES:
To evaluate the PK of YH35324 | Serum concentrations of YH35324 will be observed for 113 days after administration
  Serum concentrations of YH35324
To evaluate the PD of YH35324 | Change in serum Free/Total IgE level will be observed for 113 days after administration
  Change in serum Free/Total IgE level

OTHER OUTCOMES:
To explore the PD of YH35324 | Changes in FcεRI expression will be observed for 57days after administration
  Changes in FcεRI expression
To explore inhibition on allergens (allergy antigens) of YH35324 | Changes in allergen-induced skin prick wheal response will be observed for 57 days after administration
  Changes in allergen-induced skin prick wheal response
To explore the immunogenicity of YH35324 | Incidence of serum Anti-YH35324 antibodies will be observed for 113 Days after administration
  Incidence of serum Anti-YH35324 antibodies
To explore inhibition on allergens (allergy antigens) of YH35324 | Changes in allergen-induced serum allergen specific IgE level will be observed for 57 days after administration
  Changes in serum allergen specific IgE level

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Asan Medical Center, Pungnap-tong, Seoul
  - Severance Hospital, Yonsei University Health System, Sinchon-dong, Seoul
  - Seoul National University Bundang Hospital, Gumi, Sungnamsi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yhcho@yuhan.co.kr.
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yhcho@yuhan.co.kr.